CLINICAL TRIAL: NCT03805009
Title: Efficacy of End-Effector Robot-Assisted Gait Training in Subacute Stroke Patients: Clinical and Gait Outcomes
Brief Title: Efficacy of End-Effector Robot-Assisted Gait Training in Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 15/13
Record Dates: First submitted 2019-01-10; First posted 2019-01-15 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-06

CONDITIONS: Severe Stroke; Acute Stroke; Mild Stroke; Central Nervous System Diseases; Cerebrovascular Disease; Brain Diseases; Cardiovascular Diseases; Gait, Hemiplegic
Keywords: Stroke; Robot; Hemiparesis; Gait Training; Rehabilitation; Functional Recovery; Robot-Assisted Gait Training
MeSH Terms: conditions — Stroke; Central Nervous System Diseases; Cerebrovascular Disorders; Brain Diseases; Cardiovascular Diseases; Gait Disorders, Neurologic; Paresis

STUDY DESIGN:
Intervention Model Description: Single blinded, non randomized, pilot study
Who Masked: Outcomes Assessor
Masking Description: All the clinical assessments are routinely administered by both participating centers, and the outcome assessors are blinded to the study protocols.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Group (RG) (Experimental): Robotic Group (RG) will perform, in addition to conventional therapy, gait training using an end-effector robotic device for Robot-Assisted Gait Training (RAGT), 3 times/week for 20 sessions. During the training, patients will be asked to walk, at a varying speed, for 45 minutes and a partial Body Weight Support (BWS). Participants will start with 30-40% of BWS and an initial speed of 1.5 km/h; increasing to a maximum of between 2.2 and 2.5 km/h and reducing the initial BWS to 15%. The therapist will provide any help during sessions if required. Over 45 minutes, the patient simulates a minimum of 300 steps; patients could rest during the session, though they will be asked to walk continuously for a minimum of 5 minutes during each session.
  Interventions: Device: Robot-Assisted Gait Training (RAGT)
- Conventional Group (CG) (No Intervention): Conventional Group (CG) will perform conventional gait rehabilitation program. The treatment will include: muscle strengthening exercises and stretching of the lower limb, and static and dynamic exercises for the recovery of balance in the supine and standing positions using assistive devices; training gait exercises with parallel bars or in open spaces performed both with and without assistive devices; training to climb up and down stairs; exercises to improve proprioception in the supine, sitting and standing positions, using a proprioceptive footboard; exercises to improve trunk control.

INTERVENTIONS:
Device: Robot-Assisted Gait Training (RAGT) — The Robotic Group (RG) performs a Robot-Assisted Gait Training (RAGT) using an end-effector robotic device (G-EO system-Reha Technology-Olten, Switzerland).
  Arms: Robotic Group (RG)

SUMMARY:
To date, no studies seems to compare conventional gait rehabilitation program with end-effector RAGT in subacute stroke patients by analysing the variations of gait kinematics beyond clinical multi prospective outcomes.

The aim of this pilot study is to evaluate the efficacy of end-effector RAGT in subacute stroke patients in terms of clinical outcomes and gait kinematics, comparing them with conventional gait rehabilitation program.

DETAILED DESCRIPTION:
To evaluate the efficacy of end-effector RAGT in subacute stroke patients in terms of clinical outcomes and gait kinematics, comparing them with conventional gait rehabilitation program, patients following first ever stroke in sub-acute phase will be recruited and assessed both clinically and instrumentally (Gait Analysis) at baseline (T0) and at the end of training program (T1). The patients will be divided into 2 groups and will conduct two different types of gait training: one group will be recruited by IRCCS San Raffaele Pisana of Rome and will perform, in addition to conventional therapy, gait training using an end-effector robotic device for RAGT(Robotic Group, RG); and another group will be recruited by the Don Carlo Gnocchi Foundation Onlus of Rome, and will perform conventional gait rehabilitation program(Conventional Group, CG).

ELIGIBILITY:
Inclusion Criteria:

* first cerebral stroke
* 2 weeks up to 6 months post the acute event (subacute patients)
* age between 18-80 years
* ability to fit into the end-effector footplates
* no significant limitation of joint range of motion
* ability to tolerate upright standing for 60 seconds
* ability to walk unassisted or with little assistance
* ability to give written consent
* compliance with the study procedures

Exclusion Criteria:

* contractures of the hip, knee, or ankle joints that might limit the range of motion during gait
* medical issue that precludes full weight bearing and ambulation (e.g. orthopaedic injuries, pain, severe osteoporosis, or severe spasticity)
* cognitive and/or communicative disability (e.g. due to brain injury): inability to understand the instructions required for the study
* cardiac pathologies, anxiety or psychosis that might interfere with the use of the equipment or testing

Written informed consent was obtained from each subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-03-19 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Six-Minute Walking Test (6MWT) | Session 1 (baseline), and Session 20 (week 7)
  The 6MWT measures the distance a subject covers during an indoor gait on a flat, hard surface in 6 minutes, using assistive devices, as necessary. The test is a reliable and valid evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance. The minimal detectable change in distance for people with sub-acute stroke is 60.98 meters. The 6MWT is a patient self-paced walk test and assesses the level of functional capacity. Patients are allowed to stop and rest during the test. However, the timer does not stop. If the patient is unable to complete the test, the time is stopped at that moment. The missing time and the reason of the stop are recorded. This test will be administered while wearing a pulse oximeter to monitor heart rate and oxygen saturation, also integrated with Borg scale to assess dyspnea.

SECONDARY OUTCOMES:
Change in Fugl-Meyer Assessment (FMA) scale | Session 1 (baseline), and Session 20 (week 7)
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. The scale is comprised of five domains and there are 155 items in total:
  * Motor functioning (the score ranges from 0 (hemiplegia) to 100 points (normal motor performance). Divided into 66 points for upper extremity and 34 points for the lower extremity.
  * Sensory functioning (from 0 to 24 points)
  * Balance (from 0 to 14)
  * Joint range of motion (from 0 to 44)
  * Joint pain (from 0 to 44 ) Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.
Change in Motricity Index (MI) | Session 1 (baseline), and Session 20 (week 7)
  The MI aims to evaluate lower limb motor impairment after stroke, administrated on both sides.
  Items to assess the lower limbs are 3, scoring from 0 to 33 each: (1) ankle dorsiflexion with foot in a plantar flexed position (2) knee extension with the foot unsupported and the knee at 90° (3) hip flexion with the hip at 90° moving the knee as close as possible to the chin. (no movement: 0, palpable flicker but no movement: 9, movement but not against gravity :14, movement against gravity movement against gravity: 19, movement against resistance: 25, normal:33)
Change in Modified Ashworth Scale (MAS) | Session 1 (baseline), and Session 20 (week 7)
  The MAS is a 6 point ordinal scale used for grading hypertonia in individuals with neurological diagnoses. A score of 0 on the scale indicates no increase in tone while a score of 4 indicates rigidity. Tone is scored by passively moving the individual's limb and assessing the amount of resistance to movement felt by the examiner.
Change in Tinetti Scale Balance (TIN-B) | Session 1 (baseline), and Session 20 (week 7)
  Scales to measure activity ICF domain.
Change in Tinetti Walking (TIN-W) | Session 1 (baseline), and Session 20 (week 7)
  Scales to measure activity ICF domain.
Change in Functional Ambulation Classification (FAC) | Session 1 (baseline), and Session 20 (week 7)
  Functional Ambulation Classification is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
Change in Trunk Control Test (TCT) | Session 1 (baseline), and Session 20 (week 7)
  The TCT assesses the motor impairment in stroke patients and it's correlated with eventual walking ability. Testing is done with the patient lying on a bed: (1) roll to weak side. (2) roll to strong side. (3) balance in sitting position on the edge of the bed with the feet off the ground for at least 30. (4) sit up from lying down. Total score: 0-100
Change in 10 Meter Walk Test (10MWT) | Session 1 (baseline), and Session 20 (week 7)
  This test will assess the patient's speed during gait. Patients will be asked to walk at their preferred maximum and safe speed. Patients will be positioned 1 meter before the start line and instructed to walk 10 meters, and pass the end line approximately 1 meter after. The distance before and after the course are meant to minimize the effect of acceleration and deceleration. Time will be measured using a stopwatch and recorded to the one hundredth of a second (ex: 2.15 s). The test will be recorded 3 times, with adequate rests between them. The average of the 3 times should be recorded.
Change in Time Up And Go (TUG) | Session 1 (baseline), and Session 20 (week 7)
  The Time Up And Go is a test used to assess mobility, balance, and walking in people with balance impairments. The subject must stand up from a chair (which should not be leant against a wall), walk a distance of 3 meters, turn around, walk back to the chair and sit down - all performed as quickly and as safely as possible. Time will be measured using a chronometer.
Change in Walking Handicap Scale (WHS) | Session 1 (baseline), and Session 20 (week 7)
  The Walking Handicap Scale is a classification of 6 functional walking categories, considered as a participation category of the ICF because of its 3 items referred to community ambulation. The score ranges from 1 to 6, and do higher values represent a better outcome.

OTHER OUTCOMES:
Gait Analysis | Session 1 (baseline), and Session 20 (week 7)
  Kinematic and kinetic gait parameters will be calculated from data acquired with a motion capture system (SMART-DX; BTSBioengneering, Italy).
Postural Analysis | Session 1 (baseline), and Session 20 (week 7)
  Posturographic parameters will be obtained from the analysis of the center of pressure (COP) trajectories measured by force platforms during standing in both open and closed eyes conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Franceschini, MD, Study Chair — IRCCS San Raffaele Pisana; Sanaz Pournajaf, Dr, Principal Investigator — IRCCS San Raffaele Pisana; Michela Goffredo, Ing, Principal Investigator — IRCCS San Raffaele Pisana
Locations (2):
- Italy (2):
  - IRCCS San Raffaele Pisana, Rome, RM
  - Fondazione Don Carlo Gnocchi Onlus, Rome, RM

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Palmieri L, Barchielli A, Cesana G, de Campora E, Goldoni CA, Spolaore P, Uguccioni M, Vancheri F, Vanuzzo D, Ciccarelli P, Giampaoli S; Research Group of the Project 'Italian National Register of Coronary and Cerebrovascular Events'. The Italian register of cardiovascular diseases: attack rates and case fatality for cerebrovascular events. Cerebrovasc Dis. 2007;24(6):530-9. doi: 10.1159/000110423. Epub 2007 Oct 29. PMID 17971632
- [Background] Swinnen E, Beckwee D, Meeusen R, Baeyens JP, Kerckhofs E. Does robot-assisted gait rehabilitation improve balance in stroke patients? A systematic review. Top Stroke Rehabil. 2014 Mar-Apr;21(2):87-100. doi: 10.1310/tsr2102-87. PMID 24710969
- [Background] Eng JJ, Tang PF. Gait training strategies to optimize walking ability in people with stroke: a synthesis of the evidence. Expert Rev Neurother. 2007 Oct;7(10):1417-36. doi: 10.1586/14737175.7.10.1417. PMID 17939776
- [Background] Langhorne P, Coupar F, Pollock A. Motor recovery after stroke: a systematic review. Lancet Neurol. 2009 Aug;8(8):741-54. doi: 10.1016/S1474-4422(09)70150-4. PMID 19608100
- [Background] Mehrholz J, Thomas S, Werner C, Kugler J, Pohl M, Elsner B. Electromechanical-assisted training for walking after stroke. Cochrane Database Syst Rev. 2017 May 10;5(5):CD006185. doi: 10.1002/14651858.CD006185.pub4. PMID 28488268
- [Background] Pons, J. L. (2008). Wearable robots: biomechatronic exoskeletons. John Wiley & Sons. 127-164.
- [Background] Hesse S, Waldner A, Tomelleri C. Innovative gait robot for the repetitive practice of floor walking and stair climbing up and down in stroke patients. J Neuroeng Rehabil. 2010 Jun 28;7:30. doi: 10.1186/1743-0003-7-30. PMID 20584307
- [Background] Mehrholz J, Pohl M. Electromechanical-assisted gait training after stroke: a systematic review comparing end-effector and exoskeleton devices. J Rehabil Med. 2012 Mar;44(3):193-9. doi: 10.2340/16501977-0943. PMID 22378603
- [Background] Kelley CP, Childress J, Boake C, Noser EA. Over-ground and robotic-assisted locomotor training in adults with chronic stroke: a blinded randomized clinical trial. Disabil Rehabil Assist Technol. 2013 Mar;8(2):161-8. doi: 10.3109/17483107.2012.714052. Epub 2012 Sep 20. PMID 22992166
- [Background] Cho DY, Park SW, Lee MJ, Park DS, Kim EJ. Effects of robot-assisted gait training on the balance and gait of chronic stroke patients: focus on dependent ambulators. J Phys Ther Sci. 2015 Oct;27(10):3053-7. doi: 10.1589/jpts.27.3053. Epub 2015 Oct 30. PMID 26644642
- [Background] Li L, Ding L, Chen N, Mao Y, Huang D, Li L. Improved walking ability with wearable robot-assisted training in patients suffering chronic stroke. Biomed Mater Eng. 2015;26 Suppl 1:S329-40. doi: 10.3233/BME-151320. PMID 26406020
- [Background] Bonnyaud C, Pradon D, Boudarham J, Robertson J, Vuillerme N, Roche N. Effects of gait training using a robotic constraint (Lokomat(R)) on gait kinematics and kinetics in chronic stroke patients. J Rehabil Med. 2014 Feb;46(2):132-8. doi: 10.2340/16501977-1248. PMID 24162795
- [Background] Lonini L, Shawen N, Scanlan K, Rymer WZ, Kording KP, Jayaraman A. Accelerometry-enabled measurement of walking performance with a robotic exoskeleton: a pilot study. J Neuroeng Rehabil. 2016 Mar 31;13:35. doi: 10.1186/s12984-016-0142-9. PMID 27037035
- [Background] Gandolfi M, Geroin C, Picelli A, Munari D, Waldner A, Tamburin S, Marchioretto F, Smania N. Robot-assisted vs. sensory integration training in treating gait and balance dysfunctions in patients with multiple sclerosis: a randomized controlled trial. Front Hum Neurosci. 2014 May 22;8:318. doi: 10.3389/fnhum.2014.00318. eCollection 2014. PMID 24904361
- [Background] Sale P, Russo EF, Russo M, Masiero S, Piccione F, Calabro RS, Filoni S. Effects on mobility training and de-adaptations in subjects with Spinal Cord Injury due to a Wearable Robot: a preliminary report. BMC Neurol. 2016 Jan 28;16:12. doi: 10.1186/s12883-016-0536-0. PMID 26818847
- [Background] Dundar U, Toktas H, Solak O, Ulasli AM, Eroglu S. A comparative study of conventional physiotherapy versus robotic training combined with physiotherapy in patients with stroke. Top Stroke Rehabil. 2014 Nov-Dec;21(6):453-61. doi: 10.1310/tsr2106-453. PMID 25467393
- [Background] Hornby TG, Campbell DD, Kahn JH, Demott T, Moore JL, Roth HR. Enhanced gait-related improvements after therapist- versus robotic-assisted locomotor training in subjects with chronic stroke: a randomized controlled study. Stroke. 2008 Jun;39(6):1786-92. doi: 10.1161/STROKEAHA.107.504779. Epub 2008 May 8. PMID 18467648
- [Background] Aprile I, Iacovelli C, Padua L, Galafate D, Criscuolo S, Gabbani D, Cruciani A, Germanotta M, Di Sipio E, De Pisi F, Franceschini M. Efficacy of Robotic-Assisted Gait Training in chronic stroke patients: Preliminary results of an Italian bi-centre study. NeuroRehabilitation. 2017;41(4):775-782. doi: 10.3233/NRE-172156. PMID 28946585
- [Background] Taveggia G, Borboni A, Mule C, Villafane JH, Negrini S. Conflicting results of robot-assisted versus usual gait training during postacute rehabilitation of stroke patients: a randomized clinical trial. Int J Rehabil Res. 2016 Mar;39(1):29-35. doi: 10.1097/MRR.0000000000000137. PMID 26512928
- [Background] Mao YR, Lo WL, Lin Q, Li L, Xiao X, Raghavan P, Huang DF. The Effect of Body Weight Support Treadmill Training on Gait Recovery, Proximal Lower Limb Motor Pattern, and Balance in Patients with Subacute Stroke. Biomed Res Int. 2015;2015:175719. doi: 10.1155/2015/175719. Epub 2015 Nov 16. PMID 26649295
- [Background] Davis RB, Ounpuu S, Tyburski D, Gage JR. A gait analysis data collection and reduction technique. Hum MovSci 1991; 10: 575-587.
- [Background] Winter DA. Biomechanics and motor control of human movement. John Wiley & Sons, 2009.
- [Background] Nichols-Larsen DS, Clark PC, Zeringue A, Greenspan A, Blanton S. Factors influencing stroke survivors' quality of life during subacute recovery. Stroke. 2005 Jul;36(7):1480-4. doi: 10.1161/01.STR.0000170706.13595.4f. Epub 2005 Jun 9. PMID 15947263